CLINICAL TRIAL: NCT01829165
Title: A Causal Neural Network-level Understanding of Depression and Its Treatment Through Concurrent TMS and fMRI
Brief Title: Brain Imaging of rTMS Treatment for Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: The Dana Foundation (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Amit Etkin, Principal Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21206; P30MH089888-01 (NIH)
Record Dates: First submitted 2013-03-21; First posted 2013-04-11 (Estimated); Results first posted 2018-04-10 (Actual); Last update posted 2018-04-10 (Actual); Status verified 2018-03

CONDITIONS: Major Depressive Disorder; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- rTMS Treatment (Experimental): rTMS will be delivered for 20 sessions over 4 weeks. Active 10 Hz rTMS will be delivered using neuro-navigation based on participants' own fMRI images. Daily treatment regiments will last 36.5 minutes and rTMS will be delivered at 120% of the participant's motor threshold. Participants will be monitored during the rTMS sessions for adverse events and/or side effects.
  Interventions: Device: rTMS Treatment
- Sham Treatment (Sham Comparator): rTMS will be delivered for 20 sessions over 4 weeks. Placebo 10Hz rTMS will be delivered through sham stimulation electrodes. The rTMS coil will be positioned using neuro-navigation based on participants' own fMRI images, mimicking active rTMS treatment. Daily treatment regiments will last 36.5minutes and sham rTMS will be delivered at 120% of the participant's motor threshold. Participants will be monitored during the rTMS sham sessions for adverse events and/or side effects.
  Upon completing the sham 20 sessions participants are unblinded and offered 20 further treatments of guaranteed open-label treatment. The open-label treatment would follow the active rTMS treatment protocol.
  Interventions: Device: Sham rTMS Treatment

INTERVENTIONS:
Device: rTMS Treatment — MRI-compatible TMS stimulator
  Other Names: Magstim Stimulator; Magventure Stimulator
  Arms: rTMS Treatment
Device: Sham rTMS Treatment
  Arms: Sham Treatment

SUMMARY:
The overarching goal of this research program is to elucidate causal and directional neural network- level abnormalities in depression, and how they are modulated by an individually-tailored, circuit-directed intervention. By using concurrent TMS and fMRI, the investigators can overcome a major limitation of neuroimaging - the inability to demonstrate causality. The investigators' findings will serve as a platform for future studies wherein TMS treatment can be directly guided by the investigators' ability to image and causally manipulate specific neural networks.

Aim 1: To examine causal interactions between two major brain networks in depression.

Aim 2: To examine the impact of antidepressant TMS on causal network abnormalities in depression.

Hypothesis 1: Depressed subjects will show blunted responses, compared to healthy controls, in two targeted and interacting networks, using concurrent transcranial magnetic stimulation (TMS) and functional magnetic resonance imaging (fMRI).

Hypothesis 2: Treatment of patients with high-frequency repetitive TMS (rTMS) will result in normalization of baseline network-level deficits, and be predicted by degree of baseline network abnormalities.

DETAILED DESCRIPTION:
This study has a single primary outcome measure and other measures are exploratory. Previous versions of this study record incorrectly listed some exploratory outcome measures as secondary.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, ages 18 to 50
* Depression assessed through phone screen
* Must comprehend English well to ensure adequate comprehension of the fMRI and TMS instructions, and of clinical scales
* Has failed >1 previous adequate antidepressant medication trials
* Right-handed
* No current or history of neurological disorders
* No seizure disorder or risk of seizures

Exclusion Criteria:

* Any contraindication to being scanned in the 3T scanners at the Lucas Center or CNI such as having a pacemaker or implanted device that has not been cleared for scanning at the Lucas Center or CNI
* Any unstable medical condition, any significant CNS neurological condition such as stroke, seizure, tumor, hemorrhage, multiple sclerosis, etc
* Current rTMS treatment or prior treatment failure with rTMS
* Current electroconvulsive therapy (ECT) or prior treatment failure with ECT
* Currently pregnant or breastfeeding

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2012-09; Primary Completion 2017-01-20 (Actual); Study Completion 2017-01-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Palo Alto, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 85 participants were enrolled and 33 were randomized.
Groups:
- rTMS Treatment: Rapid transcranial magnetic stimulation (rTMS) was to be delivered for 20 sessions over 4 weeks. Active 10 Hz rTMS was delivered using neuro-navigation based on participants' own functional magnetic resonance imaging (fMRI) images. Daily treatment regiments were to last 36.5 minutes and rTMS was delivered at 120% of the participant's motor threshold. Participants were monitored during the rTMS sessions for adverse events and/or side effects.
  rTMS Treatment: MRI-compatible TMS stimulator
- Sham Treatment: Sham rTMS was to be delivered for 20 sessions over 4 weeks. Placebo 10Hz rTMS was delivered through sham stimulation electrodes. The rTMS coil was positioned using neuro-navigation based on participants' own fMRI images, mimicking active rTMS treatment. Daily treatment regiments were to 36.5minutes and sham rTMS was delivered at 120% of the participant's motor threshold. Participants were monitored during the rTMS sham sessions for adverse events and/or side effects.
  Upon completing the sham 20 sessions participants are unblinded and offered 20 further treatments of guaranteed open-label treatment. The open-label treatment would follow the active rTMS treatment protocol.
  rTMS Treatment: MRI-compatible TMS stimulator
Period: Overall Study
Arm/Group | rTMS Treatment | Sham Treatment
Started | 20 | 13
Completed | 18 | 13
Not Completed | 2 | 0
Not completed — Did not complete intervention | 2 | 0

BASELINE CHARACTERISTICS:
Population: Randomized and treated
Groups:
- rTMS Treatment: rTMS was to be delivered for 20 sessions over 4 weeks. Active 10 Hz rTMS was delivered using neuro-navigation based on participants' own fMRI images. Daily treatment regiments were to last 36.5 minutes and rTMS was delivered at 120% of the participant's motor threshold. Participants were monitored during the rTMS sessions for adverse events and/or side effects.
  rTMS Treatment: MRI-compatible TMS stimulator
- Total: Total of all reporting groups
Arm/Group | rTMS Treatment | Sham Treatment | Total
Number analyzed (Participants) | 20 | 13 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 13 | 33
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.2 (11.2) | 35.0 (6.5) | 36.2 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 20
  Male | 9 | 4 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 3 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 14 | 9 | 23
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Hamilton Depression Rating Scale (HAM-D 24) [Mean (Standard Deviation); unit: units on a scale] — The Hamilton Depression Rating Scale (HAM-D) is a 24-item clinician-administered assessment utilized as a way of determining a patient's level of depression before, during, and after treatment. Subscale scores are 0-2 (10 questions), 0-3 (2 questions), and 0-4 (12 questions). Subscales are totaled for an overall score (range 0 -76). For the overall score and all subscales, lower scores correspond to fewer symptoms, and higher scores correspond more symptoms.
  units on a scale | 27.0 (8.0) | 26.2 (5.9) | 26.9 (7.1)

OUTCOME MEASURES:

1. Primary Outcome: Clinician Administered HAM-D
Description: The Hamilton Depression Rating Scale (HAM-D) is a 24-item clinician-administered assessment utilized as a way of determining a patient's level of depression before, during, and after treatment. It takes approximately 15-20 minutes to complete the interview and score the results. Subscale scores are 0-2 (10 questions), 0-3 (2 questions), and 0-4 (12 questions). Subscales are totaled for an overall score (range 0 -76). For the overall score and all subscales, lower scores correspond to fewer symptoms, and higher scores correspond more symptoms.
Time Frame: Baseline; Day 10; Day 20
Population: Randomized and treated
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | rTMS Treatment | Sham Treatment
Number analyzed (Participants) | 20 | 13
units on a scale
  Baseline | 27.0 (8.0) | 26.2 (5.9)
  Day 10 | 22.0 (9.3) | 22.7 (6.9)
  Day 20 | 17.9 (9.9) | 17.6 (9.8)

2. Other Pre Specified Outcome: fMRI/TMS Assessed Neural Network Connectivity
Description: From pre- to post-treatment, improvement will be based on enhanced functional connectivity.
Time Frame: Up to 3 months.
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Implicit Emotion Regulation
Description: Implicit emotion regulation assessed through emotion conflict task performed during functional imaging. Performance based on reaction time and recruitment of emotion regulation regions during the task.
Time Frame: Up to 3 months
Reporting Status: Not Posted

4. Other Pre Specified Outcome: fMRI-assessed Resting Connectivity
Description: From pre- to post-treatment of patients with high-frequency repetitive TMS (rTMS) improvement shall be measured by normalization of baseline network-level deficits.
Time Frame: Up to 3 months.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 9 months
Description: Randomized and treated population
Arm/Group | rTMS Treatment | Sham Treatment
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/13
Other Adverse Events (participants affected / at risk) | 1/20 | 1/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | rTMS Treatment (N=20) | Sham Treatment (N=13)
Startled by rTMS device (Nervous system disorders) | 1 | 0
Abdominal Cramping Pain (General disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-17): https://cdn.clinicaltrials.gov/large-docs/65/NCT01829165/Prot_SAP_000.pdf